

## **Non-interventional Study Protocol**

| Document Number: | c38958167-01 |
|---|---|
| BI Study Number: | 1200-0318 |
| BI Investigational<br>Product (s): | Giotrif® (afatinib) |
| Title: | Real-world study on afatinib as first-line treatment in patients with epidermal growth factor receptor (EGFR) mutation-positive advanced non-small cell lung cancer (NSCLC) |
| Brief lay title The study observes afatinib as first-line treatment in patients with epidermal growth factor receptor (EGFF mutation-positive advanced non-small cell lung cancel.) | |
| Protocol version identifier: | 3.0 |
| Date of last version of | 26 Aug 2019 (v2.0) |
| protocol: | 03 July 2019 (v1.0) |
| PASS: | No |
| EU PAS register number: | TBD |
| Active substance: | Afatinib Antineoplastic agents, tyrosine kinase inhibitors ATC code: L01XE13 |
| Medicinal product: | Giotrif®, 30 mg and 40 mg tablets |
| Product reference: | 30 mg: EU/1/13/879/004, EU/1/13/879/005,<br>EU/1/13/879/006<br>40 mg: EU/1/13/879/007, EU/1/13/879/008,<br>EU/1/13/879/009 |
| Procedure number: | N/A |
| Joint PASS: | No |
| Research question and objectives: | Primary objective: To assess the time on treatment of afatinib as first-line therapy in advanced non-small cell lung cancer patients with EGFR mutation. Time on treatment (TOT) is defined from the start of afatinib treatment until the end of the afatinib treatment or death date by any cause. |

| | Secondary objective: |
|---|---|
| | To assess objective response rate, overall survival and safety of afatinib first-line therapy in advanced NSCLC patients with EGFR mutation. |
| | Exploratory Objective: |
| | To collect data on acquired resistance mechanism (T790M mutation, etc) to afatinib first-line therapy. |
| Country (-ies) of | China |
| study: | |
| Author: | |
| Study Team | : Clinical Trial Leader |
| Members: | |
| | : Biostatistician |
| | : Data management |
| | : Epidemiologist |
| | PV Physician |
| 35 3 4 | : Publication |
| Marketing authorisation holder: | |
| manuficial notation | |
| In case of PASS, add: | N/A |
| MAH contact person: | |
| In case of PASS, add:<br>EU-QPPV: | N/A |
| In case of PASS, add: | N/A |
| Signature of EU- | |
| QPPV: | |
| Date: | 8 Mar 2022 |

© 2022 Boehringer Ingelheim International Group of companies.All rights reserved..

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

## 1. TABLE OF CONTENTS

| TITLE PAGI | E | 1 |
|------------|--------------------------------|----|
| 1. TABLE | E OF CONTENTS | 3 |
| 2. LIST O | F ABBREVIATIONS | 6 |
| 3. RESPO | NSIBLE PARTIES | 8 |
| 4. ABSTF | RACT | 9 |
| 4.1 FLO | W CHART | 12 |
| 5. AMEN | DMENTS AND UPDATES | 15 |
| 6. MILES | TONES | 18 |
| 7. RATIO | NALE AND BACKGROUND | 19 |
| 8. RESEA | RCH QUESTION AND OBJECTIVES | 21 |
| 9. RESEA | RCH METHODS | 22 |
| 9.1 STU | DY DESIGN | 22 |
| 9.2 SET | TING | 22 |
| 9.2.1 | Study population | 23 |
| 9.2.2 | Study duration | 24 |
| 9.2.3 | Eligibility | 24 |
| 9.2.4 | Study visits | 25 |
| 9.2.5 | Study discontinuation | |
| 9.3 VAI | RIABLES | |
| 9.3.1 | Exposures | |
| 9.3.2 | Outcomes | |
| 9.3.2.1 | , | |
| 9.3.2.2 | Secondary outcomes | 28 |
| 0.2.2 | | 20 |
| 9.3.3 | Covariates | |
| | TA SOURCES TDY SIZE | |
| | TA MANAGEMENT | |
| 9.6.1 | Electronic data capture system | |
| 9.6.2 | Data entry | |
| 9.6.3 | Statistical software | |
| | TA ANALYSIS | |
| | Main analysis | 30 |

| 9.7.3 | Safety Analysis | . 31 |
|---|---|---|
| 9.8 QU | ALITY CONTROL | . 31 |
| 9.9 LIN | MITATIONS OF THE RESEARCH METHODS | . 31 |
| 9.9.1 | Lost to follow-up | . 32 |
| 9.9.2 | Channelling bias | . 32 |
| 9.9.3 | Study Sample Size | . 32 |
| 9.10 OTI | HER ASPECTS | . 32 |
| 9.10.1 | Data quality assurance | . 32 |
| 9.10.2 | Patient completion | . 33 |
| 9.10.3 | Completion of study | |
| 9.10.4 | Study records | |
| 9.10.4 | | |
| 9.10.4 | | |
| 9.10.5 | Protocol deviations | |
| 9.10.6 | Compensation available to the patient in the event of study related inju | ıry33 |
| | S 33 | |
| | ECTION OF HUMAN SUBJECTS | . 34 |
| | JDY APPROVAL, PATIENT INFORMATION, AND INFORMED NSENT | . 34 |
| | ATEMENT OF CONFIDENTIALITY | |
| | AGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE TIONS | 36 |
| | FINITIONS OF ADVERSE EVENTS | |
| | VERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION PORTING | |
| 11.3 REI | PORTING TO HEALTH AUTHORITIES | . 40 |
| | S FOR DISSEMINATING AND COMMUNICATING STUDY RESU | |
| 13. REFEI | RENCES | . 42 |
| 13.1 PUI | BLISHED REFERENCES | . 42 |
| 13.2 UN | PUBLISHED REFERENCES | . 45 |
| ANNEX 1. I | LIST OF STAND-ALONE DOCUMENTS | . 46 |
| ANNEX 2. I | ENCEPP CHECKLIST FOR STUDY PROTOCOLS | . 47 |
| ANNEX 3. A | ADDITIONAL INFORMATION | . 48 |
| ANNES 3. | 1 ECOG PERFORMANCE STATUS | . 48 |

| Boehringer Ingelheim | <b></b> |
|---|---|
| Non-interventional Study Protocol | |
| BI Study Number 1200-0318 | c38958167-01 |
| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or m | ore of its affiliated companies |
| ANNES 3.2 PROPOSED TNM STAGE GROUPINGS | 48 |
| ANNES 3.3 RECIST GUIDELINE, VERSION 1.1 | 49 |
| ANNEX 4 REVIEWERS AND APPROVAL SIGNATURES | 50 |

## 2. LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event(s)

AESI Adverse Event of Special interest ASD Absolute Standardised Differences

BI Boehringer Ingelheim
CA Competent Authority
CI Confidence Interval
CTL Clinical Trial Leader
CTM Clinical Trial Manager
CR Complete Response

CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organisation

CTCAE Common Terminology Criteria for Adverse Events

CUP Compassionate Use Programmes

DCR Disease Control Rate

EAP Expanded Access Programme eCRF Electronic Case Report Form

ECOG Eastern Cooperative Oncology Group

EDC Electronic Data Capture

EGFR Epidermal Growth Factor Receptor

EU European Union

FDA Food and Drug Administration

GCP Good Clinical Practice

GEP Good Epidemiological Practice

GPP Good Pharmacoepidemiology Practice

IB Investigator's Brochure

ICH International Conference on Harmonisation

IEC Independent Ethics Committee
IRB Institutional Review Board
ISE Institutional Review Board

ISF Investigator Site File

MAH Marketing Authorisation Holder MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Regulatory Activities

N Number

NCI National Cancer Institute
 NGS Next generation sequencing
 NIS Non-Interventional Study
 NSCLC Non-Small Cell Lung Cancer
 ORR Objective Response Rate

OS Overall Survival

PASS Post-Authorisation Safety Study

PD Progressive Disease

PFS Progression-Free Survival

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1200-0318


c38958167-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

PR Partial Response
PS Performance score
PT Preferred Term

RDC Remote Data Capture SAE Serious Adverse Event SAS Statistical Analysis Software

SD Stable Disease

SEAP Statistical and Epidemiological Analysis Plan

SmPC Summary of Product Characteristics

SOC System Organ Classes

SOP Standard Operating Procedures SqCC Squamous Cell Carcinoma

T790M Thr790Met

TKI Tyrosine Kinase Inhibitor

TMF Trial Master File TOT Time on treatment

TTF Time-to-Treatment Failure

US United States

VEGF Vascular Endothelial Growth Factor

WHO World Health Organisation

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. RESPONSIBLE PARTIES

This study is sponsored by Boehringer Ingelheim (BI).

BI appointed a clinical trial leader (CTL) who is responsible for coordinating the activities required in this study. CTL will manage the study in accordance with applicable regulations and internal standard operating procedures (SOPs). In addition, CTL will instruct the study team to conduct related procedures in this study, including preparing, conducting and reporting, ordering the materials as needed for the study. CTL will ensure that appropriate training and information are delivered to internal clinical trial manager (CTM), clinical research associates (CRAs) or external contract research organisation (CRO) members (CRO Project Managers and/or CRO CRAs), and investigators of participating sites.

The study will be done by a CRO with which the responsibilities and tasks will have been agreed and a written contract filed before initiation of the study. Data management and statistical evaluation will be performed by a CRO, which is appointed by the sponsor.

Tasks and functions assigned to organise, manage and evaluate the study will be defined according to BI SOPs. A list of responsible persons and relevant local information (as reference in protocol if applicable) are in the investigator site file (ISF) and the trial master file (TMF) document.

A coordinating investigator and a co-coordinating investigator will be nominated to coordinate principal investigators at different sites participating in this multicentre study. Tasks and responsibilities for the coordinating investigator will be defined in a contract filed before the initiation of the study.

Relevant documentation on the participating (principal) investigators and other important participants (e.g., their curricula vitae) will be filed in the ISF. An ISF containing all relevant study related documentation will be maintained according to local regulations and BI SOPs at each study site.

## 4. ABSTRACT

| Name of comp | anv: | | |
|---|---|---|---|
| Boehringer Ing | | | |
| Name of finish | | | |
| product: | | | |
| Giotrif <sup>®</sup> | | | |
| Name of active | ingredient: | | |
| Afatinib | _ | | |
| Protocol | Study | Version/Revision: | Version/Revision date: |
| date: | number: | | |
| 03 July 2019 | 1200-0318 | 3.0 | 26 Aug 2019 8 Mar 2022 |
| Title of | | on afatinib as first-line treatr | |
| study: | with EGFR muta | tion-positive advanced non-si | mall-cell lung cancer |
| Rationale | A fatinih an imax | versible ErbB family blocker, | is approved in anidarmal |
| and | | eptor-tyrosine kinase inhibito | * |
| background: | • | showed a median progressio | , |
| | • | 1.0 months in previous clinica | ` , |
| | | as first-line treatment in patie | |
| | | ll cell lung cancer (NSCLC) | |
| | | showed a significant better n | |
| | · | (TTF) versus geftinib in LUX | |
| | | LUX-Lung 6 trials, patients | · · |
| | | nths [LUX-Lung 3 OS with I | |
| | 21.1m, HR0.54(0 | 0.36-0.79), LUX-Lung 6 OS v | with Del19 patients: 31.4m |
| | vs 18.4m, HR0.64(0.44-0.94) OS benefit versus platinum-base | | |
| | chemotherapy (P15-00344). In addition, in LUX-Lung trials, afatinib | | |
| | demonstrated clinical benefit in patients with baseline brain metastases | | |
| | | ommon mutations G719X,L8 | |
| | | 2). However, resistance devel | |
| | | nmon mechanism of resistanc | |
| | ` | %) was the emergence of a s | econd-site EGFR-mutation, |
| | thr790met (T790) | M) ( <u>R15-6101</u> , <u>P09-09950</u> ). | |
| | | d real world data with afatini | |
| | | ed NSCLC Chinese patients w | |
| | | udy aims to assess the effecti | <u> </u> |
| | first-line treatment in EGRF mutated, advanced NSCLC Chinese patients | | |
| | in routine clinical | 1 | |
| Research | 1 2 3 | ective of this study is to assess | |
| question and | | ne therapy in advanced NSCl | • |
| objectives: | | on treatment (TOT) is defined | |
| | | e end of the afatinib treatmen | it or death date by any |
| | cause. | | |
| | The secondomy of | ojectives of this study are to a | ssass objective response |
| | The secondary of | ricatives of this study are to a | ccacc objective recoonce |

| Name of comp<br>Boehringer Ing<br>Name of finish<br>product:<br>Giotrif® | elheim | |
|---|---|---|
| Name of activ | e ingredient: | |
| | rate, overall survival and safety of afatinib first-line theraph NSCLC patients with EGFR mutation. The exploratory objective is to collect data on acquired remechanism (T790M mutation, etc.) to afatinib first-line the | sistance |
| Study<br>design: | Non-interventional, prospective, multicentre study based of data of Chinese EGFR-mutated NSCLC patients treated w first-line treatment. | |
| Population: | It is planned that approximately 10 study centres in China will participate in this non-interventional study (NIS), and 76 eligible patients will be enrolled. Every patient who fulfils eligibility criteria and agrees to participate in the study will be enrolled in the study. Recruitment of patients for this study is competitive. Inclusion criteria: | |
| | <ul> <li>Patients who are diagnosed with locally advanced or metastatic NSCLC with EGFR sensitive mutation</li> <li>Patients who will initiate afatinib as first-line treatment for EGFR mutation-positive NSCLC</li> <li>Male or female patients age ≥18 years</li> <li>Written informed consent per local regulatory requirement</li> </ul> | |
| | <ul> <li>Patients who have received previous systemic ther adjuvant or neo-adjuvant therapies are permitted)</li> <li>Patients with symptomatic brain metastases (patient metastases, who were previously treated, are eligible they have asymptomatic brain metastasis for at leastable doses of medication) at the start of afatinibite.</li> <li>Patients with concurrent participation in an interve Oncology clinical trial during the first-line treatment within the last 30 days prior to the first-line treatment patients join another interventional study during the second-line treatment or later-line treatment, this prior to be excluded from this study.</li> </ul> | nts with brain ble provided st 4 weeks on reatment ntional nt phase or ent phase. If e period of |
| Variables: | Primary outcomes Time on treatment of afatinib (ToT) as first-line therapy in small cell lung cancer patients with EGFR mutation. Time defined from the start of afatinib treatment until the end of treatment or death date by any cause. Patients that are lost | on treatment is the afatinib |

| Name of comp | oany: | | |
|---|---|---|---|
| Boehringer Ing | • | | |
| Name of finish | ed medicinal | | |
| product: | | | |
| Giotrif <sup>®</sup> | . in an aliant. | | |
| Name of active Afatinib | e ingreaient: | | |
| Attainio | known contact. Secondary outcome Overall survival of to follow up (inc.) Objective response according to REC Adverse events (AEs (ADRs) as in according to Uniterminology criteria. | the end of study will be censored. (OS) from the start of afatinib luding patient withdrawal) or onse rate (ORR), [objective resored complete response (CR), patients of the start of the start of afatinib first-line (CIST 1.1 with afatinib first-line (CIST), serious adverse events (INT), serious adverse events (INT) indicated by incidence, serious ted States (US) national cancer afor AEs version 5.0 (CTC). | o until the date of death, loss end of study period esponse is defined as best artial response (PR)] ne therapy (SAEs), afatinib-related sness and intensity graded er institute's (NCI) common |
| | Further outcome Resistance mecha first-line treatment | anisms (Type and proportion:<br>nt. | T790M,etc) after afatinib |
| Data | Data for this stud | ly will be obtained via the foll | lowing sources: |
| sources: | - Patient medical information: The investigator or authorized medical staff will record clinical and treatment data from patients' medical records into an electronic case report form (eCRF) at baseline and at every visit up to end of the follow up period (refer to Section 9.4) | | |
| Study size: | 76 patients | | |
| Study duration: | maximum of app collection for this | data collection for an individual<br>proximately 33 months, It is an<br>s study started from May 2020<br>il December 2023 (two years | nticipated that all data 0(first patient enrolled) and |
| Data<br>analysis: | and the median T<br>confidence interv<br>analysed similarl<br>Objective respon | nt (TOT) will be analysed using time on Treatment (TOT) along al (CI) will be calculated. Over y. se rate (ORR) and acquired remarised descriptively by frequency. | ng with two-sided 90%<br>erall survival (OS) will be<br>esistance mutation type, and |
| Milestones:<br>IRB/IEC Appro<br>First Patient In | oval: May 2020<br>: May 2020 | | |

| Name of company: |
|----------------------------|
| Boehringer Ingelheim |
| Name of finished medicinal |
| product: |
| Giotrif <sup>®</sup> |
| Name of active ingredient: |
| Afatinib |
| Last Patient In: Dec 2021 |
| Interim Analysis: Dec 2022 |
| Last Patient Out: Dec 2023 |
| Database Locked: Mar 2024 |
| Final NIS Report: Jun 2024 |

## 4.1 FLOW CHART

## **Table 1. Patient Flow Chart**

| Procedure | Baseline | Treatment (first-line) | Treatment (second-line) | Further<br>subsequent<br>treatment(s)<br>up to death | End of<br>study<br>(Until Dec<br>2023 or<br>death) |
|---|---|---|---|---|---|
| Observation period | Before initiation of afatinib | Initiation of afatinib first-line treatment: Followed by regular visits according to institution standards | Start second-<br>line treatment<br>(first visit ≤1<br>months<br>followed by<br>regular visits<br>according to<br>institution<br>standards) | Start further subsequent treatment(s) followed by regular visits according to institution standards | |
| Informed consent <sup>a</sup> | X | | | | |
| Demographics (age, gender, height, etc.) | X | | | | |
| Body weight | X | X | | | |
| Presence of brain metastases | X | X | | | |
| Afatinib dose | | X | | | |
| ECOG Performance Status | X | X | | | |
| Baseline characteristics Type of EGFR mutation at start of afatinib therapy Genetic testing information Disease stage Comorbidities | Xª | | | | |

| Medical history | | | | | |
|---|---|---|---|---|---|
| Laboratory testing information <sup>c</sup> | X | X | | | |
| Eligibility (I/E criteria) | X | | | | |
| Administration/Concomitant therapies | X | X | X | | |
| Tumour assessment<br>according to local<br>institutional standards <sup>d</sup> | X | X | X | | |
| Patient vital status | X | X | X | X | X |
| Regular follow-up | | X | X | | |
| Genetic testing <sup>b</sup> | | | X <sup>f</sup> | | |
| Adverse events (AEs) | X | X | Xe | Xe | Xe |

<sup>&</sup>lt;sup>a</sup>: Written informed consent must be obtained before any screening/baseline data collection are performed.

f: Genetic testing is needed according to clinical practice prior to subsequent treatment.

b: Genetic testing report (including PCR, NGS, etc.) will be collected if available

<sup>°:</sup> Detailed Laboratory tests are included in <u>section 9.3.3</u>. The estimated GFR (glomerular filtration rate) using modification of diet in renal disease (MDRD) formula, eGFR = 186 x SCr (mg/dL)<sup>-1.154</sup> x Age<sup>-0.203</sup> x (0.742 if female) (<u>R02-2529</u>).

d: Tumour assessment will only be applied while patients with anti-tumour therapy (first-line and second-line or later lines). If the treatment finish, the assessment will end.

<sup>&</sup>lt;sup>e:</sup> All AEs have to be collected and documented on the eCRF from the day of signing informed consent up to 30 days after the last dose of afatinib administration. In addition, all ADRs associated with afatinib and AEs with fatal outcome must be collected and documented on the eCRF after the end of residual effect period (30 days after the last dose of afatinib administration) up to the end of study. Progression of underlying malignancy is exempted from reporting as adverse event on the eCRF AE page and on the NIS AE form, when considered not related to afatinib, requirements for reporting on NIS AE form are included in section 11.2.

## Below Firure 1 is the study flow chart:

## Figure 1:Study Flow Chart



Prospective Data collection

(patients enrollment period : 2020 May – 2021 Dec) Demographics (age, gender, height, body weight, etc.)

· Baseline characteristics

Type of EGFR mutation at start of afatinib therapy Genetic testing information

Disease stage

Comorbidities

Medical history

Presence of brain metastases

ECOG Performance Status

- Laboratory testing information
- · Administration/Concomitant therapies
- · Patient vital status

Prospective Data collection

(patients follow up period:2020 May-2022 Dec)

- Date of afatinib last dose
- Afatinib dose
- Adverse events & AE leading to dose modification
- Genetic testing after <u>afatinib</u> first-line failure ( if applicable)
- Subsequent therapy medication (after <u>afatinib</u> first-line therapy failure)
- · Presence of brain metastases
- ECOG Performance Status
- · Patient vital status
- · Date of Death

Expected Outcomes: TOT, ORR, Safety,

Prospective Data collection

(patients follow up period:2022 Dec-2023 Dec)

- Date of afatinib last dose
- Afatinib dose
- Adverse events & AE leading to dose modification
- Genetic testing after <u>afatinib</u> first-line failure (if applicable)
- Subsequent therapy medication (after afatinib first-line therapy failure)
- · Presence of brain metastases
- ECOG Performance Status
- · Patient vital status
- · Date of Death

Expected Outcomes :OS, updated TOT

## 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1.0 | 03<br>Jul<br>2019 | NA | NA NA | NA |
| 2.0 | 26<br>Aug<br>2019 | Refer to<br>Protocol<br>Version 2.0 | Refer to Protocol version 2.0 | Refer to<br>Protocol<br>Version 2.0 |

| 3.0 | 8<br>Mar<br>2022 | 4 | Abstract updating per protocol 3.0 | Abstract updating per protocol 3.0 |
|---|---|---|---|---|
| | | 6 | Milestone updating per updated study timeline | Milestone<br>updating per<br>updated study<br>timeline |
| | | 7 | Adding related information of study rationale and background: 1. Afatnib clinical benefit in uncommon EGFR mutation and brain metastases. 2. Limited real world data with afatinib first-line treatment in EGFR-mutated, advanced nonsmall cell lung cancer Chinese patients. | Study rationale<br>and<br>background<br>changing |
| | | 8 | Primary objective and secondary objective were updated to: 1. The primary objective of this study is to assess the time on treatment of afatinib as first-line therapy in advanced non-small cell lung cancer patients with EGFR mutation. Time on treatment (TOT) is defined from the start of afatinib treatment until the end of the afatinib treatment 2. The secondary objective is to assess objective response rate, overall survival and safety of | Research<br>question and<br>objectives<br>updating per<br>study rationale |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| afatinib first-line therapy in advanced NSCLC patients with EGFR mutation. To collect data on acquired resistance mechanism (T790M mutation, etc) to afatinib first-line therapy. | |
|---|---|
| Related sessions in research methods were updated to: 1. Study design: This NIS will be conducted at 10 study sties in China and the patients treated with first-line afatinib will be followed up until death, lost to follow-up, withdraw from the study, or end of the study for other reasons, whichever comes first and no later than 2023. 2. Study Setting: 76 patients treated with afatinib first line treatment, will be enrolled into this prospective NIS across multiple centres in China. 3. Study Variables - Outcomes: Primary outcome is time on treatment of afatinib as first-line therapy in advanced non-small cell lung cancer patients with EGFR mutation. Time on Treatment (TOT) is defined from the start of afatinib treatment until the end of the afatinib treatment. Patients that are lost to follow up or withdraw before the end of study will be censored at the time of last known contact. Secondary outcomes are overall survival, Objective response rate, Resistance mechanisms and safety. 4. Study size: Seventy-six patients will be included in this study. 5. Data analysis: We conducted time on treatment (TOT) of afatinib first-line therapy and overall survival (OS) for the main analysis. Moreover, ORR, | Research methods updating per updated study objectives |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | resistance mechanism and AEs will be for further analysis. If data allows, it would also be of interest to look at the overall survival in patients who had different subsequent treatments after afatinib. | |
|---|---|---|
| 11 | Updating Adverse events reporting with Pregnancy | Updating Adverse events reporting with Pregnancy |

## 6. MILESTONES

| Milestone | Planned Date |
|------------------|--------------|
| IRB/IEC Approval | May 2020 |
| First Patient In | May 2020 |
| Last Patient In | Dec 2021 |
| Interim Analysis | Dec 2022 |
| Last Patient Out | Dec 2023 |
| Database Locked | Mar 2024 |
| Final NIS Report | Jun 2024 |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RATIONALE AND BACKGROUND

Lung cancer is the leading cause of cancer-associated mortality worldwide. In 2018, World Health Organisation (WHO) reported approximately 2.1 million new lung cancer cases annually and 1.8 million deaths which represents 18.4% of the total cancer deaths worldwide (R18-3308). In China, lung cancer is also considered as a leading cause of death among males. A total of 0.73 million new lung cancer cases and 0.61 million deaths (R18-1649). For NSCLC, it accounts for approximately 85% of all primary lung cancers where most patients were presented with advanced and unresectable disease at the time of diagnosis (R18-3355, R08-2617).

Current available therapeutic strategy varies depending on the disease stages with some combining local treatments (surgery and/or radiotherapy) and systemic treatments (chemotherapy and/or targeted therapy). Systemic therapies are the mainstay treatment for patients with stage IIIb/IV (unresectable cancers) (P11-07424). These may include chemotherapy, vascular endothelial growth factor (VEGF) inhibitor, immunotherapy and target therapy. Treatment with EGFR-TKI is the preferred option for patients with EGFR gene mutation as metastatic EGFR-mutant lung cancers are sensitive to EGFR TKIs (P18-01881).

Acquired resistance to EGFR-targeted TKIs therapy is inevitable due to tumour evolution. Kohsaka and team reported in 2018 that EGFR mutation-positive NSCLC is highly heterogeneous at the cellular level, facilitating clonal expansion of resistant tumours via multiple molecular mechanisms (<u>P18-10855</u>). To date, the 6 approved EGFR-TKIs can be classified into three different generations - 1st generation (erlotinib, gefitinib and icotinib), 2nd generation (afatinib and dacomitinib) and 3rd generation (osimertinib) (<u>R18-0130</u>, <u>P19-03609</u>).

Efficacy and safety of TKIs of different generation are widely investigated in WJTOG3405, NEJ002, ARCHER 1050, EURTAC, OPTIMAL, NEJ026, LUX-Lung 3, LUX-Lung 6, LUX-Lung 7, AURA3 and FLAURA(P19-00432). The range of PFS reported with the longest being 18.9 months was indicated in patients who were with EGFR-mutated advanced NSCLC and treated with osimertinib as the first-line (FLAURA) comparing to standard of care (10.2 months) (either received gefitinib or erlotinib) in EGFR mutant NSCLC treatment naïve patients (R18-0130). To date, osimertinib it is the only commercially approved 3rd generation EGFR TKI for the treatment of patients with EGFR thr790met (T790M) positive tumour in China (P19-00432).

The first marketing authorisation of afatinib was granted on 12 Jul 2013 in the US (trade name Gilotrif®) as first-line treatment for patients with metastatic NSCLC and whose tumours have EGFR exon 19 deletions or exon 21 (L858R) substitution mutations as detected by an FDA-approved test (P13-10659) and the indication was updated in 2018 in US for the First-line treatment of patients with metastatic non-small cell lung cancer (NSCLC) whose tumours have non-resistant EGFR mutations as detected by an FDA-approved test. In the European Union (EU), afatinib was approved on 25 Sep 2013 (trade name Giotrif®) as monotherapy for the treatment of EGFR TKI-naïve patients with locally advanced or metastatic NSCLC with activating EGFR mutation(s). Furthermore, in US and EMA, afatinib is also approved in for squamous cell carcinoma (SqCC) of the lung progressing after

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

platinum-based chemotherapy. In China, afatinib (trade name Giotrif<sup>®</sup>) was approved on 21 Feb 2017 for patients with NSCLC with activating EGFR mutation that previously were not treated with EGFR TKI and for squamous cell carcinoma (SqCC) of the lung progressing after platinum-based chemotherapy.

Afatinib showed a median PFS of approximately 11 months in treatment-naïve patients with EGFR common and uncommon mutations in LUX-Lung 3 (P13-07382), LUX-Lung 6 (P14-00758) and LUX-Lung 7 (P16-04350). Furthermore, when comparing with gefitinib, it reduced the risk of PFS (HR=0.73 [95% CI 0·57–0·95],) in LUX-Lung 7. In addition, in LUX-Lung trials, afatinib demonstrated clinical benefit in patients with baseline brain metastases and with the uncommon mutations G719X,L861Q, and S768I (P16-01306,P15-05932). Nevertheless, most patients (approximately >50%) developed resistance to either 1st or 2nd generation EGFR TKIs due to the emergence of a second-site EGFR-mutation, the T790M (R15-6101, P09-09950).

There are limited real world data with afatinib first-line therapy in EGFR-mutated, advanced non-small cell lung cancer Chinese patients who are treatment naive. Therefore, this study aims to assess the effectiveness and safety of afatinib first-line treatment in EGFR mutated, advanced non-small cell lung cancer Chinese patients in routine clinical practice.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. RESEARCH QUESTION AND OBJECTIVES

Data from real-world setting will provide information on afatinib first-line treatment in Chinese patients diagnosed with advanced EGFR mutation-positive NSCLC.

## **Primary objective:**

• The primary objective of this study is to assess the time on treatment of afatinib as first-line therapy in advanced non-small cell lung cancer patients with EGFR mutation. Time on treatment (TOT) is defined from the start of afatinib treatment until the end of the afatinib treatment or death date by any cause. Patients that are lost to follow up or withdraw before the end of study will be censored at the time of last known contact..

#### **Secondary objective:**

• To assess objective response rate, overall survival and safety of afatinib first-line therapy in advanced NSCLC patients with EGFR mutation.

## **Exploratory objective:**

To collect data on acquired resistance mechanism (T790M mutation, etc) to afatinib first-line therapy.

## 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This is a NIS to be conducted at approximately 10 sites in China where real world data are from EGFR mutation positive NSCLC patients who will initiate afatinib as first-line treatment and receiving subsequent therapy. All the study sites will need to have afatinib used in regular clinical practice. Participating investigators will screen patients for eligibility, obtain informed consent, and enrol patients who meet the eligibility criteria. Investigators or trained site personnel will then complete the eCRF to capture information on demographic, medical history, and treatment information at the time of enrolment.

This study will only include patients who are newly diagnosed and who will receive afatinib as first-line treatment, regardless if they will receive 3rd generation or other treatment subsequently. Data will be collected for the patients who receiving afatinib first-line therapy and subsequent therapy. Data of patients' resistance mechanism after afatinib treatment will also be collected.

Day 0 is the date that the patient sign the informed consent. Day 1 is the first dose of afatinib. We collected the date of initial and metastatic diagnosis. Day 1 is the first dose of afatinib therapy (index date). The patients will be followed up by regular visits according to institution standards after start of afatinib until death, lost to follow-up, withdraw from the study, or end of the study for other reasons, whichever comes first and no later than Dec 2023. Please refer to Section 4.1 for the visit plan and major information collected during each visit.

This study is descriptive only and there are no comparisons between groups. To assess the presence of this bias (discussed in Section 9.9), data from 1200.0066 study [where patients were diagnosed with locally advanced or metastatic NSCLC harbouring EGFR mutation(s)] may be used to verify if this study contains potential channelling bias.

#### 9.2 SETTING

76 patients, who are diagnosed with locally advanced or metastatic NSCLC (with activating EGFR mutation) and will be treated with afatinib as fist line treatment, are be enrolled into this prospective NIS across multiple centres in China.

Eligibility will be assessed prior to enrolment during a scheduled visit. Patients who fulfil eligibility criteria as well as agree to participate in the study by signing an informed consent (required by local regulation and legal requirement) will be included into the study.

Participation of patients in this study is not intended to change the routine treatment that patients receive as determined by their clinicians; all treatment decisions, type and timing of disease monitoring are at the discretion of the treating physician. Patients will be followed by regular visits according to institution standards after the treatment is initiated. Study sites

Site selection criteria in China:

- Sites prescribe afatinib on a regular clinic basis to patients with EGFR mutationpositive NSCLC
- Capability of conducting an NIS, including qualification, experience, availability and research resource of investigators
- A genetic test [(next-generation sequencing (NGS) or polymerase chain reaction, (PCR)] is applicable for patients diagnosed with NSCLC

After completing the sites feasibility for this study, 10 study sites participated in this prospective observational study.

**Table 2. Study Sites** 

| No | City | Site |
|----|-----------|------|
| 1 | Beijing | |
| 2 | Chengdu | |
| 3 | Zhengzhou | |
| 4 | Hangzhou | |
| 5 | Haikou | |
| 6 | Zhongshan | |
| 7 | Guangzhou | |
| 8 | Guangzhou | |
| 9 | Shenyang | |
| 10 | Shenzhen | |

## 9.2.1 Study population

Eligible patients will be enrolled in this study and will receive afatinib (first-line) and subsequent treatment (second-line) of either 3rd generation EGFR TKI or other treatments.

Patients who are administrated with a fatinib as first-line treatment started from May 2020 (first patient enrolled) and will be followed up until death, lost to follow-up, withdraw from

the study, or end of the study for other reasons, whichever comes first and no later than Dec 2023.

#### 9.2.2 Study duration

It is anticipated that all data collection for this study started from May 2020 (first patient enrolled) and will continue until Dec 2023 or the event of OS. The maximum duration of data collection for an individual patient will be a maximum of 33 months. this period may be truncated due to treatment switching, patient withdrawal from the study, or death or end of study for any other reason.

#### 9.2.3 Eligibility

Patients must meet all of the following inclusion criteria and not meet any of the exclusion criteria to be eligible for the study:

#### • Inclusion criteria:

- o Patients who are diagnosed with locally advanced or metastatic NSCLC with EGFR sensitive mutation positive
- Patients who will initiate afatinib as first-line treatment for EGFR mutation-positive NSCLC
- Male and female patients with age  $\ge$ 18 years
- Written informed consent per local regulatory requirement

#### • Exclusion criteria:

- Patients who have received previous systemic therapy (previous adjuvant or neo-adjuvant therapies are permitted)
- O Patients with symptomatic brain metastases (patients with brain metastases, who were previously treated, are eligible provided they have asymptomatic brain metastasis for at least 4 weeks on stable doses of medication) at the start of afatinib treatment
- Patients with concurrent participation in an interventional oncology clinical trial during the first-line treatment phase or within the last 30 days prior to the first-line treatment phase. If patients join another interventional study during the period of second-line treatment or later-line treatment, this patient should not be excluded from this study

All patients who fulfil eligibility criteria and provide written informed consent will be enrolled

Patients' record in the study will be maintained in the ISF at the investigational sites.

## 9.2.4 Study visits

This NIS does not impose a therapy protocol, diagnostic/therapeutic procedure, but a regular clinical visit schedule. Patients will be enrolled in the study during a regularly scheduled clinic visit prior to initiating their treatment (Day 0). Day 1 is defined as the day that the patient initiates afatinib (index date). Patients will be followed by regular visits according to institution standards since enrolment. After progression on first-line treatment with afatinib, based on the clinical practice, patients may have an appropriate genetic examination (such as NGS or PCR) in order to identify the best treatment option based on the testing result.

Lab testing and additional procedures would be based on physician's judgement and clinical practice.

Below Figure 1 list the study flow chart and visits

Figure 1: Study Flow Chart



## 9.2.5 Study discontinuation

BI reserves the right to discontinue the study or at a particular study site at any time for the following reasons:

- Failure to meet expected enrolment goals overall or at a particular study site
- Emergence of any efficacy/safety information that could significantly affect the continuation of the study, or any other administrative reasons

• Violation of regulations, the study protocol, or the contract by a study site, disturbing the appropriate conduct of the study

The investigator/the study site will be reimbursed for reasonable expenses incurred in the event of study termination (except in the event of the third reason).

#### 9.3 VARIABLES

This is a prospective, observational study. Clinical data will being collected and enters data directly into the eCRF during or after the patient visit per study protocol. The study protocol does not mandate treatments, each participating site provides and documents patient care and outcomes according to usual care, physician discretion and local practice standards. Thus, study variables may not be available for all patients at all data collection time points per routine medical care. All the data will be continuously and directly into the eCRF during or after the patient visit in the whole study period.

The study variables to be collected include:

- Date of diagnosis
- Demographics: age at the start of afatinib treatment, gender, smoking status
- Laboratory test: hematology, biochemistry and urine examinations. List below table 2:

Table 3. Laboratory test

| Category | Parameters |
|---|---|
| Hematology | Hemoglobin, platelet count, white blood cell (WBC), absolute neutrophil count (ANC) |
| Chemistry | Electrolytes: Sodium and potassium Liver function tests: Alkaline phosphatase, aspartate amino transferase (AST/SGOT), alanine amino transferase (ALT/SGPT), γ-glutamyltransferase (GGT), total bilirubin Renal function parameters: Blood urea/Blood Urea Nitrogen (BUN), creatinine |
| | Other: Glucose, albumin, phosphorus, lactate dehydrogenase (LDH), total protein, |
| Urinalysis | pH, protein, glucose, blood/erythrocytes, leucocytes, nitrite; in case of clinically significant finding further evaluation should be performed and results documented. Dipstick testing is sufficient. |

- Stage of disease at the start of afatinib treatment
- Tumour histology

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Type of EGFR mutations at the start of afatinib and subsequent treatment, specifically the type of acquired resistance mutation
- Sites of metastases at start of afatinib treatment
- Body weight and height at the start of afatinib treatment
- Eastern cooperative oncology group (ECOG) performance score (PS) (if available) at start of afatinib treatment
- Date of start and end of afatinib treatment
- Starting dose of afatinib
- Afatinib dose modification(s) and date(s) (if applicable)
- ECOG PS (if available) at start of subsequent treatment
- Sites of metastases at the start of subsequent treatment
- Reason for discontinuation of afatinib treatment (e.g., progressive disease (PD), AE)
- If subsequent treatment was provided within an expanded access programme (EAP)/compassionate use programmes (CUP) or prescribed as clinical practice
- Comorbidities (hepatitis B, gastritis, liver cirrhosis, etc.)
- Concomitant medications including (PPIetc.)
- AEs (leading to dose modification)
- Date & Cause of death

## 9.3.1 Exposures

#### Afatinib:

Patients will be treated with afatinib 30 mg or 40 mg tablet once daily as indicated in the approved labels of afatinib.

## 3rd generation EGFR TKI or other subsequent treatment:

Patients may be treated with 3rd generation EGFR TKI or other subsequent treatment as indicated in the approved labels.

The Summaries of Product Characteristics on Giotrif® is contained in the ISF in the "Summary of Product Characteristics" (SmPC) section.

#### 9.3.2 Outcomes

## 9.3.2.1 Primary outcomes

Time on treatment of afatinib as first-line therapy in advanced non-small cell lung cancer patients with EGFR mutation. Time on Treatment (TOT) is defined from the start of afatinib treatment until the end of the afatinib treatment. Patients that are lost to follow up or withdraw before the end of study will be censored at the time of last known contact.

#### 9.3.2.2 Secondary outcomes

- Overall Survival(OS) from the start of afatinib until the end of study, date of death, patient withdrawal or loss to follow-up
- ORR [OR is defined as best overall response of CR and PR] according to RECIST 1.1 by investigator review with afatinib in first-line treatment
- AEs, SAEs, afatinib-related AEs (ADRs) as indicated by incidence seriousness and intensity graded according to United States (US) national cancer institute's (NCI) (CTCAE Version 5.0)



#### 9.3.3 Covariates

As mentioned previously, the data from study 1200-0066 will be used to assess presence of potential channelling bias and to put the results into perspective. Therefore, the baseline characteristics of patients in 1200-0066 trial will be described. The covariates to be collected in the both studies (if applicable) are listed as following.

- Baseline demographic: age, gender, height, weight, body mass index, , smoking status (former, current, never)
- Clinical characteristics including medical history, surgery history, lab testing information (haematology, biochemistry and urine examinations), disease stage, tumour histological classification, EGFR mutation at start of afatinib therapy, ECOG PS score, brain metastases, afatinib starting dose
- Current/Concomitant medications

#### 9.4 DATA SOURCES

Data for this study will be obtained via the following sources:

- Patient medical information: The investigator or authorised medical staff will record clinical and treatment data from patients' medical records/laboratory tests/physical examination into an eCRF at baseline and at every visit up to the end of the follow-up period.

There are no protocol-mandated tests, procedures, or clinic visits for this study. All the data will be continuously and directly into the eCRF during or after the patient visit in the whole study period.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.5 STUDY SIZE

Seventy-six patients will be included in this study.

Based on LUX-Lung trials, we assume the median time on treatment (TOT) on afatinib to be 12 months in this study. Assuming that the time on treatment (TOT) follows an exponential distribution, it is expected to have 35 events till 2 years after last patient in, given total sample size equal to 76, considering a 30% drop out rate.

#### 9.6 DATA MANAGEMENT

#### 9.6.1 Electronic data capture system

Data will be gathered in the electronic data capture (EDC) system prepared by the sponsor or appointed CRO. The details of data management procedures to ensure the quality of the data will be described in the statistical and epidemiological analysis plan (SEAP) available in eTMF.

#### 9.6.2 Data entry

All the data will be continuously and directly into the eCRF during or after the patient visit in the whole study period. All reported data from the enrolled investigator's site will be entered via a secured web-based EDC study database. All site personnel will be fully trained in using the EDC system, including eCRF completion guidelines. Site personnel will be provided with secure usernames and passwords in order to enter study data into the EDC system. All participating sites will only have access to view and enter the data for their patients. A data manager will perform concurrent review during the course of the data collection period. Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The Investigator may need to request previous medical records or transfer records, depending on the study; also current medical records must be available. For eCRFs all data must be derived from source documents. Data queries generated from the database will be created on an ongoing basis, queries will be based on the data management system logic deck and database validation for adequacy and consistency. The site management team will follow-up to request the completion of such queries.

#### 9.6.3 Statistical software

All analyses will be performed using statistical analysis software (SAS) for Microsoft Windows operating system statistical software (version 9.3 or higher, using validated implementations of each application or SAS custom programming.

#### 9.7 DATA ANALYSIS

For the purpose of this study, analyses will generally be descriptive in nature and will be conducted using SAS statistical software (version 9.3 or higher). Descriptive data regarding patient demographic and clinical characteristics will be calculated. For categorical measures, data will include the frequency (number of cases (n)) and percentage (%) of total study

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

patients observed in each category (N). All variables will be summarised descriptively through tabular displays of mean, median, ranges and standard deviations of continuous variables and frequency distributions of categorical variables. When necessary, continuous variables also will be categorised into intervals, with the distribution of patients (n, N, %) for each interval provided.

AEs will be graded in accordance with CTCAE Version 5.0. The safety analyses include frequency and intensity of AEs, SAEs and ADRs by System Organ Class (SOC)/Preferred Term (PT) using a current medical dictionary for regulatory activities (MedDRA) dictionary. In addition, AEs resulting in the discontinuation of treatment will be studied.

To assess the presence of channelling bias, we will use the data from study 1200-0066 to assess potential channelling and to put the results into perspective. The baseline characteristics of patients in this study and in study 1200-0066 separately. Patient characteristics will be compared between the two groups using absolute standardised differences (ASD), where an ASD of at least 10% will be considered a meaningful difference.

## 9.7.1 Main analysis

All patients treated with afatinib will be included in the analysis of the primary outcome, Time on Treatment (TOT) on afatinib. Time on Treatment (TOT) will be evaluated by Kaplan-Meier analysis. Median Time on Treatment (TOT) and two-side 90% CI, and the quartiles will be calculated from the Kaplan-Meier curve. Patients who are lost to follow up without providing the end date of treatment with afatinib will be censored at the time of last known contact.

Overall survival (OS) will be evaluated by Kaplan-Meier analysis. Median overall survival (OS) and two-side 90% CI, and the quartiles will be calculated from the Kaplan-Meier curve. Patients who are lost to follow up (including patient withdrawal) without providing the end date of treatment will be censored at the time of last known contact. Patients who reach the end of study period without providing the end date of treatment will be censored at the end of study.



#### 9.7.3 Safety Analysis

All adverse events and adverse drug reactions collected per study protocol will be included and summarised in the interim safety analysis and in the final study report.

#### 9.8 QUALITY CONTROL

This NIS will be conducted according to Guidelines for Good Pharmacoepidemiology SPractice (GPP) and Good Pharmacovigilance Practice (GVP), and also will be conducted following the standards of International Council for Harmonisation/Good Clinical Practice (ICH/GCP) (7) in accordance with local regulations, particularly regarding ethics, protection of patient's privacy, and processing of data. All necessary related data and documents will be made available for inspection.

All entries in the eCRFs will be stored in a database. The structure of the database is based on the division into sections and entry fields defined in the eCRFs. To improve and ensure data quality, data checks will be performed automatically in the eCRFs directly on electronic entry at the study site.

Plausible value ranges for numerical data entries, and logical data and list entries will be filed in the eCRFs. The tests for consistency and completeness based on this will be performed during entry in the eCRFs. The validity of the recorded data will, therefore, be ensured by the validations incorporated in the documentation system, which highlight incorrect or implausible entries to the data entry clerk/doctor.

If corrections are necessary after the data are saved, these will be documented in an audit trail.

For further quality assurance of the documented patient observations, a sample-size based source data verification will be performed on about 30% of patients included (not including the additional data collected for follow-up analyses). In addition, a risk-based monitoring will be taken for critical data and documents of all patients, and 100% of these critical data and documents will be verified.

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by independent ethics committees (IECs) or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

Prospective data collection brings its own challenges. Even with a careful controlled design, there may be various sources of bias that can completely distort the results. In this study, potential limitations of the study design can be listed as:

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.9.1 Lost to follow-up

All patients will be followed up until the event of OS. If a patient misses more than 1 clinic care visit, the site will attempt to communicate with the patient and document the patient's reason for not returning. Sites will be requested to contact patients at various times of the day and evening and on different days of the week. If the patient cannot be contacted after the due diligence process, the treating physician will attempt to contact the patient's designated secondary contacts, including the patient's general practitioner and next-of-kin or out-of-household contacts to obtain information on the patient's whereabouts and vital status. If the patient's care has been transferred to another healthcare professional, the treating physician at the enrolling site will be responsible for obtaining the required follow-up information from the new treating physician. Patients who do not return for at least 2 scheduled visits, and for whom no information is available will be considered lost to follow-up and will be censored at time of last visit or last known contact with the healthcare provider. Follow-up information collecting could be accepted by phone call if the information is available and complete.

## 9.9.2 Channelling bias

Channelling bias can occur due to preferential prescribing in relation to different risks for the events of interest. For example, if aftinib therapy would be prescribed more often compared with other treatments to high risky Chinese patients with EGFR mutation positive NSCLC (e.g., patients in this study are more severe than other Chinese EGFR mutation positive NSCLC patients or with more comorbidities at baseline). Thus, more incidences of outcome events were expected in the group with afatinib therapy (e.g., the incidence rates of AEs/ADRs will be affected). Furthermore, all patients who fulfil eligibility criteria and provide written informed consent will be enrolled, as patients with severe disease or other disabilities (eg those who are likely to have poorer outcomes) may be excluded from the study. This study is descriptive only and there are no comparisons between groups. To assess the presence of the bias, we plan to use the data from study 1200-0066 to put the results into perspective to compare baseline demographic and clinical characteristics of the NSCLC patients. Through this, we can verify that safety or efficacy difference is due to patient baseline characteristics or the sequential therapy.

## 9.9.3 Study Sample Size

76 patients were enrolled in this study, this is a small sample size which may impact the assessment of study outcomes. A sample size of 76 patients is expected to ensure an 80% chance to observe the width of the 90% CI of median TOT of afatinib smaller than or equal to 11 months.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

#### 9.10.2 Patient completion

The collection of the data of patients will continue until the end of data collection or withdrawal of consent (if applicable) which occurs first.

## 9.10.3 Completion of study

The end of the study will occur when the data is collected from the last patient's data. No further data will be collected afterwards.

## 9.10.4 Study records

eCRFs for individual patients will be provided by the sponsor via remote data capture.

#### 9.10.4.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported on the eCRFs that are transcribed from source documents must be consistent with the source documents, or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study; also current medical records must be available.

#### 9.10.4.2 Direct access to source data and documents

The investigator/institution will permit study-related monitoring, audits, IEC review, and regulatory inspection, providing direct access to all related source data/documents. eCRFs and all source documents, including progress notes and copies of laboratory and medical test results, must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities (e.g.,NMPA). The CRA/CTM and auditor may review all eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 9.10.4.1.

#### 9.10.5 Protocol deviations

NA

#### 9.10.6 Compensation available to the patient in the event of study related injury

NA

#### **9.11 BIAS**

Methodological efforts have been taken to minimise channelling bias and attrition bias: these efforts including using the data from study 1200-0066 to assess potential channelling and to put the results into perspective, which will help address this issue. Details of bias can be referred to Section 9.9.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonised Tripartite Guideline for GCP (to the extent applicable to the NIS setting and required by local regulations), Good Epidemiological Practice (GEP), guidelines for GPP, and relevant BI SOPs. Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

## 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective IEC and competent authority (CA) according to national and international regulations. The same applies to the implementation of changes introduced by amendments.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements. Each signature must be personally dated by each signatory and the informed consent and any additional patient information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her study-related data will be used by BI in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his/her medical records may be examined by authorized monitors (CTM/CRA) or quality medicine auditors appointed by BI, by appropriate IEC members, and by inspectors from regulatory authorities.

#### 10.2 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential, and disclosure to third parties is prohibited with the exceptions noted below. Patient privacy will be ensured by using patient identification code numbers.

Data protection and data security measures are implemented for the collection, storage, and processing of patient data by principle 6 and 12 of the WHO GCP handbook.

Data generated as a result of the study need to be available for inspection on request by the participating investigators, the sponsor's representatives, by the IEC and the regulatory authorities.

## Boehringer Ingelheim Non-interventional Study Protocol BI Study Number 1200-0318


c38958167-01

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IEC and the regulatory authorities.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITIONS OF ADVERSE EVENTS

#### **Adverse event**

AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (e.g., an abnormal test finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### **Adverse reaction**

An adverse reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility. Adverse reactions may arise from the use of the product within or outside the terms of the marketing authorisation or from occupational exposure. Conditions of use outside the marketing authorisation include offlabel use, overdose, misuse, abuse, and medication errors.

## Serious adverse event

SAE is defined as any AE which

- results in death
- is life-threatening
- requires in-patient hospitalisation, or prolongation of existing hospitalisation
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly/birth defect

Life-threatening in this context refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious events, such as important medical events that might not be immediately life-threatening or result in death or hospitalisation but may jeopardise the patient or might require intervention to prevent one of the other outcomes listed above.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of drug dependency or drug abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction

Adverse Event of Special Interest (AESI)

No AESIs have been defined for this study.
## 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

The investigator shall maintain and keep detailed records of all AEs in their patient files.

## **Collection of AEs**

The study design is of non-interventional nature, and the study is conducted within the conditions of the approved marketing authorisation. Sufficient data from controlled interventional trials are available to support the evidence on the safety and efficacy of the afatinib. For this reason, the following AE collection and reporting requirements have been defined.

The following must be collected by the investigator in the eCRF from signing the informed consent onwards until the end of the study:

- From signing the informed consent onwards until 30 days after the last dose of afatinib administration:
  - \*All AEs (serious and non-serious)
- From the end of the residual effect period (30 days after the last dose of afatinib administration) onwards until the individual patient's end of study:
  - o All ADRs (serious and non-serious) associated with afatinib
  - o \*All AEs with fatal outcome

"Progressive Disease (PD) of the malignancy" is the study endpoint and will be recorded on the appropriate page of the eCRF.

During the whole study, progression of the malignancy under study (including signs and symptoms of progression) should not be reported as adverse event unless the progression is considered related to a fatinib.

When there is evidence suggesting a causal relationship between afatinib and the progression of the underlying malignancy, the event must be reported as an AE on the eCRF and on the NIS AE Form.

All AEs that are to be collectedincluding those persisting after study completion, must be followed up until they are resolved, have been sufficiently characterised, or no further information can be obtained.

#### Causal relationship of adverse event

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an AE. An adverse reaction, in contrast to an AE, is characterised by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

<sup>\*</sup>Exemption regarding progression of underlying malignancy:

Medical judgment should be used to determine the relationship, considering all relevant factors, including the pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases, and relevant history.

Arguments that may suggest a reasonable causal relationship could be:

- The event is **consistent with the known pharmacology** of the drug
- The event is known to be caused by or attributed to the drug class
- A plausible time to onset of the event relative to the time of drug exposure
- Evidence that the **event is reproducible** when the drug is re-introduced
- No medically sound alternative etiologies that could explain the event (e.g., preexisting or concomitant diseases, or co-medications)
- The event is typically **drug-related and infrequent in the general population** not exposed to drugs (e.g., Stevens-Johnson syndrome)
- An indication of dose-response (i.e., greater effect size if the dose is increased, smaller effect size if the dose is diminished)

Arguments that may suggest that there is **no reasonable possibility of a causal relationship** could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g., pre-treatment cases, diagnosis of cancer or chronic disease within days/weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into account the pharmacological properties of the compound (e.g., after 5 half-lives). Of note, this criterion may not apply to events whose time course is prolonged despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g., situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

#### Intensity of adverse event

The intensity of AEs should be classified and recorded according to the CTCAE criteria in the eCRF.

#### **Pregnancy:**

In rare cases, pregnancy might occur in a NIS. Once a patient has been enrolled in the study and has taken study medication, the investigator must report any drug exposure during pregnancy in a study participant within 7 days by means of Part A of the Pregnancy Monitoring Form to the sponsor's unique entry point.

Similarly, potential drug exposure during pregnancy must be reported if a partner of a male

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

trial participant becomes pregnant. This requires a written consent of the pregnant partner. The ISF will contain the trial specific information and consent for the pregnant partner.

The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported to the sponsor's unique entry point on the Pregnancy Monitoring Form (Part B).

The ISF will contain the Pregnancy Monitoring Form (Part A and B). As pregnancy itself is not to be reported as an AE, in the absence of an accompanying serious ADR and/or AESI, only the Pregnancy Monitoring Form and not the NIS AE form is to be completed. If there is a serious ADR and/or AESI associated with the pregnancy a NIS AE form must be completed in addition.

#### Expedited reporting of AEs and drug exposure during pregnancy

The following must be reported by the investigator on the NIS AE form and/or Pregnancy Monitoring Form from signing the informed consent onwards until the end of the study and provide o BI unique entry point:

Table 4: Expedited reporting of AEs and drug exposure during pregnancy

| Type of Report | Timeline |
|---|---|
| All <b>serious ADRs</b> associated with <del>afatinib</del> Giotrif® | immediately within 24 hours |
| All <b>AEs with fatal outcome</b> in patients exposed to afatinib Giotrif® *Exemption applies | immediately within 24 hours |
| All <b>non-serious ADRs</b> associated with afatinib Giotrif® | 7 calendar days |
| Drug exposure during pregnancy | 7 calendar days |

<sup>\*</sup>Exemption

Death due to disease progression of the underlying malignancy is a study endpoint and the natural course of the disease. As such it is exempted from reporting as an SAE. Progression of the subject's underlying malignancy will be recorded on the appropriate pages of the eCRF only and will not be reported on the NIS AE Form. However, when there is evidence suggesting a causal relationship between afatinib and the progression of the underlying malignancy, the event must be reported as an SAE on the NIS AE Form and on the eCRF.

The same timelines apply if follow-up information becomes available for the respective events. In specific occasions, the investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax and/or email the NIS AE form.

#### **Information required**

For each reportable AE, the investigator should provide the information requested on the appropriate eCRF pages and the NIS AE form (if applicable).

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 11.3 REPORTING TO HEALTH AUTHORITIES

AE reporting to regulatory agencies will be done by the Marketing Authorisation Holder (MAH) according to local and international regulatory requirements.

Exemptions are described in <u>section 11.2</u>, if applicable.

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and the sponsor with regard to the publication of the results of this study are described in the investigator contract.

The publication for study design is planned for Dec 2019, the interim analysis for the primary outcome and some secondary outcomes is planned for Dec 2022, and the publication kick-off for primary outcome is planned for Jun 2023 after the interim analysis report is completed. The final publication will be written after the final NIS report is completed in Dec 2024.

BI intends to use data from this study to prepare peer-reviewed publications and other scientific communications such as abstracts, posters, and podiums presentations.

## 13. REFERENCES

## 13.1 PUBLISHED REFERENCES

| R18-3308 | Freddie Bray, Jacques Ferlay, Isabelle Soerjomataram, et al. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. |
|---|---|
| R18-1649 | |
| | Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, et al. Cancer statistics in China, 2015. CA; 2016; 66(2); 115-132. |
| R08-2617 | Molina JR, Yang P, Cassivi SD, Schild SE, Adjei AA. Non-small cell lung cancer: epidemiology, risk factors, treatment, and survivorship. Mayo Clin Proc; 2008; 83(5); 584-594. |
| P09-09950 | Nguyen KSH, Kobayashi S, Costa DB. Acquired resistance to epidermal growth factor receptor tyrosine kinase inhibitors in non-small-cell lung cancers dependent on the epidermal growth factor receptor pathway. Clin Lung Cancer. 2009. 10 (4): 281 – 289. |
| P11-07424 | Ramalingam SS, Owonikoko TK, Khuri FR. Lung cancer: new biological insights and recent therapeutic advances. CA Cancer J clin. 2011. 61 (2): 91 - 112. |
| P13-07382 | Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, et al. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013. 31 (27): 3327 – 3334. |
| P13-10659 | Dungo RT and Keating GM. Afatinib: first global approval. Drugs 2013. 73 (13): 1503 – 1515. |
| P14-00758 | Wu YL, Zhou C, Hu CP, Feng J, Lu S, Huang Y, et al. Afatinib versus cisplatin plus gemcitabine for first-line treatment of Asian patients with advanced non-small-cell lung cancer harbouring EGFR mutations (LUX-Lung 6): an open-label, randomised phase 3 trial. Lancet Oncol. 2014. 15 (2): 213 – 222. |
| P15-11024 | Niederst MJ, Hu H, Mulvey HE, Lockerman EL, Garcia AR, Piotrowska Z, et al.The allelic context of the C797S mutation acquired upon treatment with third-generation EGFR inhibitors impacts sensitivity to subsequent treatment strategies. Clin Cancer Res. 2015. 21 (17): 3924 – 3933. |

| P15-00344 | James Chih-Hsin Yang*, Yi-Long Wu*, Martin Schuler, Martin Sebastian, Sanjay Popat, Nobuyuki Yamamoto, Caicun Zhou, et al. Afatinib versus cisplatin-based chemotherapy for EGFR mutation-positive lung adenocarcinoma (LUX-Lung 3 and LUX-Lung 6): analysis of overall survival data from two randomised, phase 3 trials. Lancet Oncol 2015; 16: 141-51. |
|---|---|
| P15-05932 | James C-H Yang*, Lecia V Sequist*, Sarayut Lucien Geater, Chun-Ming Tsai, Tony Shu Kam Mok,et al. Clinical activity of afatinib in patients with advanced non-small-cell lung cancer harbouring uncommon EGFR mutations: a combined post-hoc analysis of LUX-Lung 2,LUX-Lung 3, and LUX-Lung 6.Lancet Oncology 2015;16:7 830-838. |
| P16-01306 | Martin Schuler, MD,* Yi-Long Wu, MD, Vera Hirsh, MD, Kenneth O'Byrne, MD, et al. First-Line Afatinib versus Chemotherapy in Patients with Non–Small Cell Lung Cancer and Common Epidermal Growth Factor Receptor Gene Mutations and Brain Metastases. Journal of Thoracic Oncology. 2016 Mar;11(3):380-90. |
| P16-04350 | Park K, Tan EH, O'Byrne K, Zhang L, Boyer M, Mok T et.al. EGFR mutation-positive non-small-cell lung cancer (LUX-Lung 7): a phase 2B, open-label, randomised controlled trial. Lancet Oncol. 2016. 17 (5): 577 – 589. |
| P17-01744 | Paz-Ares L, Tan EH, O'Byrne K, Zhang L, Hirsh V, Boyer M, et al. Afatinib versus gefitinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: overall survival data from the phase IIb LUX-Lung 7 trial. Ann Oncol. 2017. 28 (2): 270 – 277. |
| P18-01881 | Arriola E, Garcia Gomez R, Diz P, Majem M, Martinez Aguillo M, Valdivia J, et al. Clinical management and outcome of patients with advanced NSCLC carrying EGFR mutations in Spain. BMC Cancer. 2018. 18 (1): 106. |
| P18-09968 | Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JCH, et al. Sequential treatment with afatinib and osimertinib in patients with EGFR mutation-positive non-small-cell lung cancer: an observational study. Future Oncol 2018.14 (27): 2861 – 2874. |
| P18-10855 | Kohsaka S, Petronczki M, Solca F, Maemondo M. Tumor clonality and resistance mechanisms in EGFR mutation-positive non-small-cell lung cancer: implications for therapeutic sequencing. Future Oncol. 2019. 15 (6): 637 – 652. |

| P18-11537 | Hochmair MJ, Morabito A, Hao D, Yang CT, Soo RA, Yang JCH, et al. Afatinib followed by osimertinib in patients with EGFR mutation-positive advanced NSCLC: a real-world study (GioTag). ESMO Asia 2018, 4th Asian Cong of the European Society for Medical Oncology (ESMO), Singapore, 23 - 25 Nov 2018 Ann Oncol. 2018. 29 (Suppl 9), IX176 - IX177, Abstr LBA7. |
|---|---|
| P19-00432 | Takeda M, Nakagawa K. First- and second-generation EGFR-TKIs are all replaced to osimertinib in chemo-naive EGFR mutation-positive non-small cell lung cancer? Int J Mol Sci. 2019.20 (1): 146. |
| P19-01037 | Hochmair M, Cufer T, Morabito A, Hao D, Yang C, Soo R, et al. Sequential treatment with afatinib and osimertinib in real-world patients with EGFR mutation-positive advanced NSCLC: the GioTag study. BTOG 2019, 17th Ann Conf of the British Thoracic Oncology Group (BTOG), Dublin, 23 - 25 Jan 2019. Lung Cancer (Neth). 2019. 127 (Suppl 1), S37, Abstr 86. |
| P19-03125 | Park K, Bennouna J, Boyer M, Hida T, Hirsh V, Kato T, et al. Sequencing of therapy following first-line afatinib in patients with EGFR mutation-positive non-small cell lung cancer. Lung Cancer (Neth). 2019. 132:126 – 131. |
| P19-03609 | Chinese Society of Lung Cancer, Chinese Anti-Cancer Association,<br>Lu S. EGFR-TKI ADR management Chinese expert consensus.<br>(Original in Chinese). Chin J Lung Cancer 2019. 22 (2): 57 – 81. |
| R02-2529 | Bosch JP, Lewis JB, Greene T, Rogers N, Roth D, et. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Ann Intern Med 1999. 130(6):461-470 |
| R15-6101 | Arcila ME, Oxnard GR, Nafa K, Riely GJ, Solomon SB, Zakowski MF, et al. Rebiopsy of lung cancer patients with acquired resistance to EGFR inhibitors and enhanced detection of the T790M mutation using a locked nucleic acid-based assay. Clin Cancer Res. 2011. 17 (5): 1169 – 1180. |
| R16-1552 | Thress KS, Paweletz CP, Felip E, Cho BC, Stetson D, Dougherty B, et al. Acquired EGFR C797S mutation mediates resistance to AZD9291 in non-small cell lung cancer harboring EGFR T790M. Nature Med. 2015. 21 (6): 560 – 562. |
| R18-0130 | Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, et al. FLAURA Investigators Osimertinib in untreated EGFR-mutated advanced non-small-cell lung cancer. N Engl J Med. 2018. 378 (2): 113 – 125. |

| R18-3355 | Brahmer JR, Govindan R, Anders RA, Antonia SJ, Sagorsky S, Davies MJ, et al. The Society for Immunotherapy of Cancer consensus statement on immunotherapy for the treatment of non-small cell lung cancer (NSCLC). J Immunother Cancer 2018. 6 (1): 75. |
|---|---|
| R09-0262 | Eisenhauer EA,et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1) Eur J Cancer; 2009; 45; 228-247. |

## 13.2 UNPUBLISHED REFERENCES

| c01617169-07 | Investigator's Brochure (IB): Afatinib (BIBW 2992), Indication: Oral Treatment of Cancer, 1200.P1/1200.P2/1200.P3/1200.P4/1200.P5/1200.P6/1200.P7/1200. P8/1200.P9/1200.P10/1200.P11/1200.P12/1200.P13/1200.P14 Version 20, 14 December 2018 |
|---|---|
| c01802941-10 | Investigator's Brochure (IB): Afatinib (BIBW 2992), Indication: Oral Treatment of Cancer,1200.P1/1200.P2/1200.P3/1200.P4/1200.P5/1200.P6/1200.P 7/1200.P8/1200.P9/1200.P10, Version 16, 06 Jul 2015 |
| c14668275-03 | Protocol for non-interventional studies: GioTag: Real-world data study on sequential therapy with Gi(l)otrif®/afatinib as first-line treatment followed by osimertinib in patients with EGFR mutation positive advanced non-small cell lung cancer |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|---|---|---|---|
| 1 | NA | 3-Sep-2019 | Informed consent form |
| 2 | NA | 26-Dec-2019 | Statistical and epidemiological analysis plan |

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Not applicable

## **ANNEX 3. ADDITIONAL INFORMATION**

## **ANNES 3.1 ECOG PERFORMANCE STATUS**

| Grade | Definition |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2 | Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4 | Completely disabled, cannot carry on any self-care, totally confined to bed or chair |
| 5 | Dead |

## **ANNES 3.2 PROPOSED TNM STAGE GROUPINGS**

| Occult carcinoma | TX | NO NO | MO |
|-----------------------|---------|-----------|-----|
| Stage 0 | Tis | NO | MO |
| Stage IA1 | T1a(mi) | NO | MO |
| | T1a | NO | MO |
| Stage IA2 | T1b | NO | MO |
| Stage IA3 | T1c | NO | MO |
| Stage IB | T2a | NO NO | MO |
| Stage IIA | T2b | NO | MO |
| Stage IIB | T1a-c | N1 | MO |
| | T2a | N1 | MO |
| | T2b | N1 | MO |
| | T3 | NO | MO |
| Stage IIIA | T1a-c | <u>N2</u> | MO |
| | T2a-b | N2 | MO |
| | T3 | N1 | MO |
| | T4 | NO | MO |
| | T4 | N1 | MO |
| Stage IIIB | T1a-c | N3 | MO |
| | T2a-b | N3 | MO |
| | T3 | N2 | MO |
| | T4 | N2 | MO |
| Stage IIIC | T3 | N3 | MO |
| Account of the second | T4 | N3 | MO |
| Stage IVA | Any T | Any N | M1a |
| | Any T | Any N | M1b |
| Stage IVB | Any T | Any N | M1c |



**ANNES 3.3 RECIST GUIDELINE, VERSION 1.1** 

Refer to the Revised RECIST guideline (version 1.1) which was published in by Eisenhauer EA,et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1) Eur J Cancer; 2009; 45; 228-247.(R09-0262)

| Target lesions | Non-target lesions | New<br>lesions | Overall<br>response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or<br>not all evaluated | No | PR |
| SD | Non-PD or<br>not all evaluated | No | SD |
| Not all<br>evaluated | Non-PD | No | NE |
| PD | Any | Yes or No | PD |
| Any | PD | Yes or No | PD |
| Any | Any | Yes | PD |

| Non-target lesio | ns N | ew lesions | Overa | ll resp | onse |
|---|---|---|---|---|---|
| CR | 3 | No | CR | | |
| Non-CR/non-PD | | No | Non-CR/non-PD | | n-PD* |
| Not all evaluated | | No | NE | | |
| Unequivocal PD | | Yes or No | PD | | |
| Any | | Yes | PD | | |
| CR = complete : NE = inevaluable. | response, | PD = progressiv | e dis | ease, | and |

## ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI<br>product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM Market<br>Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | | | |
| Global PVWG Chair | X | | |
| GPV SC | | | |
| Global CTIS representative | | | |
| Local Medical Director /Market<br>Access | X (if local study) | | X |
| Local Head MAcc / HEOR Director | | | |
| Global TA Head Epi* | | | |
| Global TA Head Clinical<br>Development / Medical Affairs /<br>Market Access* | | | |
| Global TA Head PV RM* | | | |
| RWE CoE<br>(for NISnd only) | X | X | X |
| PSTAT / PSTAT-MA<br>(for NISnd only) | X | X | X |
| NIS DM | | | |
| Local Head MA/Clinical Development | | | |

<sup>\*</sup> After review by Global TM for function

**Study Title:** Real-world study afatinib as first-line treatment in patients with epidermal growth factor receptor (EGFR) mutation-positive advanced non-small cell lung cancer (NSCLC)**Study** 

Number: 1200.0318

Protocol Version: V3. 0

I here with certify that I agree to the content of the study protocol and to all documents referenced in the study protocol.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |